CLINICAL TRIAL: NCT01839292
Title: A Newly Designed Conformable Uncovered Versus Covered Self-expandable Metallic Stent for Palliation of Malignant Gastric Outlet Obstruction: a Prospective, Randomized Multicenter Study
Brief Title: ComVi and D-type Stent in Malignant GOO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Collaborators: National Cancer Center, Korea (Other Government); Kyungpook National University Hospital (Other); Hallym University (Other); The Catholic University of Korea (Other); Seoul National University (Other); DongGuk University (Other)
Responsible Party: Principal Investigator, Sun Gyo Lim, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AJIRB-DEV-DE4-10-009
Record Dates: First submitted 2013-04-18; First posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Gastric Outlet Obstruction
Keywords: gastric outlet obstruction; palliative treatment; stent
MeSH Terms: conditions — Gastric Outlet Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- uncovered D-type stent (Active Comparator): uncovered D-type stent, which effectively reduces stent migration, especially in malignant colorectal obstruction
  Interventions: Device: uncovered D-type stent insertion
- double-layered ComVi stent (Active Comparator): double-layered ComVi stent, which is a modified covered stent with an additional outer bare wire mesh to overcome both tumor ingrowth and stent migration
  Interventions: Device: double-layered ComVi stent insertion

INTERVENTIONS:
Device: uncovered D-type stent insertion
  Arms: uncovered D-type stent
Device: double-layered ComVi stent insertion
  Arms: double-layered ComVi stent

SUMMARY:
Covered self-expandable metallic stents (SEMS) have been used to prevent tumor ingrowth, a common complication of uncovered SEMSs. However, they have revealed a high incidence of stent migration in patients with unresectable malignant gastric outlet obstruction (GOO). A conformable covered SEMS was introduced to overcome both stent migration and tumor ingrowth. The aims of this study were to evaluate the clinical outcomes of newly designed conformable covered and uncovered SEMS for palliation of malignant GOO.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 years of age or older
* obstructive symptoms due to unresectable malignant GOO
* a Karnofsky performance score of more than 30 (13)

Exclusion Criteria:

* history of a previous SEMS insertion
* the presence of obstruction in the gastrointestinal tract excluding the gastric outlet
* severe comorbidities precluding the endoscopic procedure, such as cardiopulmonary disease, sepsis, and bleeding disorders
* a life expectancy of less than 1 month after SEMS insertion
* history of gastric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
the stent patency time from stent insertion to restenosis due to stent malfunction or death | Up to 1 years

SECONDARY OUTCOMES:
stent malfunction (e.g., stent migration or occlusion due to tumor ingrowth/overgrowth) and the reintervention rate | up to 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Jin Hong Kim, M.D., Ph.D., Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, South Korea